CLINICAL TRIAL: NCT01552668
Title: The Effect of a Twice Daily, 200 mg Dose of Oral Fidaxomicin Compared to Placebo on Risk of Acquiring C. Difficile and Developing C. Difficile Infection (CDI) in High Risk Patients
Brief Title: Fidaxomicin to Prevent Clostridium Difficile Colonization
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study not performed
Sponsor: Washington University School of Medicine (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201109037; 1U54CK000162 (NIH)
Record Dates: First submitted 2012-03-08; First posted 2012-03-13 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile infection; fidaxomicin
MeSH Terms: conditions — Clostridium Infections | interventions — Fidaxomicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fidaxomicin (Experimental): Receive 200 mg of fidaxomicin twice daily
  Interventions: Drug: Fidaxomicin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fidaxomicin — Receive 200 mg of fidaxomicin twice daily
  Other Names: Dificid
  Arms: Fidaxomicin
Drug: Placebo — Receive Placebo twice daily
  Arms: Placebo

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of an antibiotic called fidaxomicin in preventing C. difficile infection.

DETAILED DESCRIPTION:
A novel approach to prevent C. difficile infection is to use compounds with activity against C. difficile as primary prophylaxis in high risk patients. Chemoprophylaxis theoretically can prevent C. difficile infection by two mechanisms. It may reduce transmission from asymptomatic C. difficile carriers by reducing the number of spores shed in the stool and prevent replication and subsequent toxin production of the organisms in patients at risk for C. difficile infection.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* On broad spectrum antimicrobials
* Anticipated length of stay of > 48 hours after enrollment
* A non-ICU inpatient

Exclusion Criteria:

* Pregnant
* Expected to die within 7 days
* Have previously been enrolled in this trial or a trial of an investigational agent to treat CDI, and/or are on monotherapy with an antimicrobial generally considered not to increase the risk of CDI (vanc, macrolides, tetracyclines, trimethoprim/sulfamethoxazole, aminoglycosides, colistin, linezolid, nitrofurantoin, metronidazole)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Clostridium difficile | At discharge from hospital (average of 7 days after enrollment in study)
  Clostridium difficile isolated from patient stool specimen

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Belmares J, Johnson S, Parada JP, Olson MM, Clabots CR, Bettin KM, Peterson LR, Gerding DN. Molecular epidemiology of Clostridium difficile over the course of 10 years in a tertiary care hospital. Clin Infect Dis. 2009 Oct 15;49(8):1141-7. doi: 10.1086/605638. PMID 19780659
- [Background] Dubberke ER. The A, B, BI, and Cs of Clostridium difficile. Clin Infect Dis. 2009 Oct 15;49(8):1148-52. doi: 10.1086/605639. No abstract available. PMID 19780660
- [Background] Bobo LD, Dubberke ER. Recognition and prevention of hospital-associated enteric infections in the intensive care unit. Crit Care Med. 2010 Aug;38(8 Suppl):S324-34. doi: 10.1097/CCM.0b013e3181e69f05. PMID 20647790
- [Background] Dubberke ER, Butler AM, Hota B, Khan YM, Mangino JE, Mayer J, Popovich KJ, Stevenson KB, Yokoe DS, McDonald LC, Jernigan J, Fraser VJ; Prevention Epicenters Program from the Centers for Disease Control and Prevention. Multicenter study of the impact of community-onset Clostridium difficile infection on surveillance for C. difficile infection. Infect Control Hosp Epidemiol. 2009 Jun;30(6):518-25. doi: 10.1086/597380. PMID 19419269
- [Background] Dubberke ER, Butler AM, Reske KA, Agniel D, Olsen MA, D'Angelo G, McDonald LC, Fraser VJ. Attributable outcomes of endemic Clostridium difficile-associated disease in nonsurgical patients. Emerg Infect Dis. 2008 Jul;14(7):1031-8. doi: 10.3201/eid1407.070867. PMID 18598621
- [Background] Dubberke ER, Butler AM, Yokoe DS, Mayer J, Hota B, Mangino JE, Khan YM, Popovich KJ, Stevenson KB, McDonald LC, Olsen MA, Fraser VJ; Prevention Epicenters Program of the Centers for Disease Control and Prevention. Multicenter study of surveillance for hospital-onset Clostridium difficile infection by the use of ICD-9-CM diagnosis codes. Infect Control Hosp Epidemiol. 2010 Mar;31(3):262-8. doi: 10.1086/650447. PMID 20100085
- [Background] Dubberke ER, Gerding DN, Classen D, Arias KM, Podgorny K, Anderson DJ, Burstin H, Calfee DP, Coffin SE, Fraser V, Griffin FA, Gross P, Kaye KS, Klompas M, Lo E, Marschall J, Mermel LA, Nicolle L, Pegues DA, Perl TM, Saint S, Salgado CD, Weinstein RA, Wise R, Yokoe DS. Strategies to prevent clostridium difficile infections in acute care hospitals. Infect Control Hosp Epidemiol. 2008 Oct;29 Suppl 1:S81-92. doi: 10.1086/591065. No abstract available. PMID 18840091
- [Background] Dubberke ER, McMullen KM, Mayfield JL, Reske KA, Georgantopoulos P, Warren DK, Fraser VJ. Hospital-associated Clostridium difficile infection: is it necessary to track community-onset disease? Infect Control Hosp Epidemiol. 2009 Apr;30(4):332-7. doi: 10.1086/596604. PMID 19239377
- [Background] Dubberke ER, Reske KA, Noble-Wang J, Thompson A, Killgore G, Mayfield J, Camins B, Woeltje K, McDonald JR, McDonald LC, Fraser VJ. Prevalence of Clostridium difficile environmental contamination and strain variability in multiple health care facilities. Am J Infect Control. 2007 Jun;35(5):315-8. doi: 10.1016/j.ajic.2006.12.006. PMID 17577478
- [Background] Dubberke ER, Reske KA, Olsen MA, McMullen KM, Mayfield JL, McDonald LC, Fraser VJ. Evaluation of Clostridium difficile-associated disease pressure as a risk factor for C difficile-associated disease. Arch Intern Med. 2007 May 28;167(10):1092-7. doi: 10.1001/archinte.167.10.1092. PMID 17533213
- [Background] Dubberke ER, Wertheimer AI. Review of current literature on the economic burden of Clostridium difficile infection. Infect Control Hosp Epidemiol. 2009 Jan;30(1):57-66. doi: 10.1086/592981. PMID 19049438
- [Background] Louie T, Miller M, Donskey C, Mullane K, Goldstein EJ. Clinical outcomes, safety, and pharmacokinetics of OPT-80 in a phase 2 trial with patients with Clostridium difficile infection. Antimicrob Agents Chemother. 2009 Jan;53(1):223-8. doi: 10.1128/AAC.01442-07. Epub 2008 Oct 27. PMID 18955525
- [Background] Louie TJ, Miller MA, Mullane KM, Weiss K, Lentnek A, Golan Y, Gorbach S, Sears P, Shue YK; OPT-80-003 Clinical Study Group. Fidaxomicin versus vancomycin for Clostridium difficile infection. N Engl J Med. 2011 Feb 3;364(5):422-31. doi: 10.1056/NEJMoa0910812. PMID 21288078